CLINICAL TRIAL: NCT05862870
Title: Mobile Application Treatment for TMD: Feasibility Trial
Brief Title: TMD Online Program for Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Mark Litt, Professor, UConn Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-052-1; 3U01DE028520-03S1 (NIH)
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: TMD/Orofacial Pain

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- painTRAINER pain management web application (Experimental): This is a patient-administered pain management training program delivered in 10 sessions over 8 weeks. Each session is composed of different skills useful for managing chronic pain. Each session is also accompanied by recommendations for skills practice to be done between sessions.
  Interventions: Behavioral: painTRAINER

INTERVENTIONS:
Behavioral: painTRAINER — patient self-administered pain management web application

SUMMARY:
This is a proposal for an administrative supplement to the parent study, "Individualized Assessment and Treatment Program for TMD: Coping as a Mechanism" (U01 DE028520). The parent study is currently engaged in exploring the extent to which the training of coping skills per se is an important mechanism of psychosocial treatment. The current project seeks to lay the groundwork for expanding the range of treatment mechanisms examined to include therapeutic relationship factors (therapist support, empathy, acknowledgment). The present supplemental study will provide instruction for individual patient pain management via an online application, with no therapist or counselor assistance. The aim is to determine the extent to which treatment-related outcomes (including adherence and pain) may be influenced by therapist support factors.

DETAILED DESCRIPTION:
Psychosocial treatments have been effective for temporomandibular disorders (TMD), but the mechanisms of action for these treatments are unclear. Most studies of psychosocial treatment, including the parent U01, have focused on relatively specific psychosocial mechanisms, including coping skills acquisition, pain management self-efficacy, decrease in catastrophizing, increased mindfulness, acceptance, and readiness to change behavior to ameliorate pain. The 2 therapist-delivered treatments in the parent study are packaged CBT or Individualized Assessment and Treatment (IATP). Left untested in this study are common therapeutic factors that often emerge as influential in pain outcome research. These common, non-specific therapeutic factors include (especially): the therapeutic alliance; interpretation and understanding; emotional expression; reinforcement; information; and reassurance and support. Because both conditions of the parent U01 involve similar levels of therapist involvement, therapist support and other treatment-non-specific variables cannot be tested clearly. One way to assess these factors is to introduce a pain treatment that explicitly does not contain these factors; i.e., a treatment that does not employ therapists or require supervision by health care professionals. There are currently no studies published in which therapist-led treatments have been compared to a mobile application-based treatment.

The Investigators therefore propose to pilot test a mobile application treatment condition (painTrainer©) added as an additional treatment condition to the parent study, and provided to 20 patients in the coming year. This condition will deliver the content of the CBT condition of the parent study, but will do so with no therapist contact. If this mobile application is found credible and acceptable it may be used in additional comparisons with treatments conducted by therapists. Thus at some point it will be possible to parse the effects of cognitive-behavioral treatment content per se and therapist support factors.

An additional benefit of testing such a mobile application is that it might in the future provide a means to expand the reach of pain management professionals to remote and underserved populations.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years
* Complaint of either bilateral or unilateral pain, scoring > 3 on a 11-point pain scale (scored from 0 to 10), in the area of the temporomandibular joint
* Pain has persisted for a period of at least 3 months by patient self-report. Pain may be constant or intermittent.

Exclusion Criteria:

* Contraindications to TMD treatment (as determined by the consulting oral surgeon)
* Inadequate fluency in English
* History of prior surgery for TMD
* Receiving concurrent treatment for orofacial pain (including orthodontic or physical therapy)
* Have a condition that requires the use of an oral appliance (e.g., sleep apnea)
* Diagnosed as having pain of neuropathic or odontogenic origin
* History of rheumatoid disease or autoimmune disease (e.g., rheumatoid arthritis; lupus) currently being treated with anti-inflammatory drugs
* History of kidney disease or current kidney issues
* Extensive anatomical destruction or deterioration of the TM joint
* Current treatment of chronic pain issue with anti-inflammatories (e.g., Indomethacin; methotrexate; dexamethasone) or opioid analgesics
* Carrying a diagnosis of psychosis (as per self-report on Quick Screen)
* Pregnant or anticipating pregnancy (due to prescription of NSAIDs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Litt, PhD, Principal Investigator — UConn Heatlh
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Summary data will be made available to interested investigators by the PI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21 persons with TMD/orofacial pain of at least 3mo duration were recruited through advertisements and referrals from local dentists
Period: Overall Study
Arm/Group | painTRAINER Pain Management Web Application
Started | 21
Completed | 18 (of 21 enrolled, 18 completed protocol)
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: We recruited 1 person more than initially planned in order to make up for losses to follow-up
Arm/Group | painTRAINER Pain Management Web Application
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Demographics: Race
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 18
    More than one race | 0
    Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 21
Graded Chronic Pain Scale [Mean (Standard Deviation); unit: units on a scale] — The Graded Chronic Pain Scale is a multidimensional measure that assesses 2 dimensions of overall chronic pain severity: pain intensity and pain-related disability. In the current study 3 items were averaged to produce a reliable pain index as an outcome measure: current pain, average pain, and worst pain in the past week
  units on a scale | 5.17 (2.02)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Feasibility
Description: Treatment is deemed feasible if 20 persons are recruited with 8 months and complete the program.
  This number of patients recruited over this time period would indicate that the program is attractive to the target patient population.
  If this number finish the program, it would indicate that the program was a feasible means of intervention.
Time Frame: 8 months
Population: 21 persons were recruited, supporting treatment feasibility
Measure: Count of Participants; unit: Participants
Arm/Group | painTRAINER Pain Management Web Application
Number analyzed (Participants) | 21
Participants | 18
Statistical Analysis 1: Comparison: painTRAINER Pain Management Web Application; Frequency count of patients retained in treatment; Test type: Other — Frequency count; p = .05, count; exact count = 20, 0% CI 2-sided [20 to 20], Standard Deviation 0.0; Threshold for frequency count

2. Primary Outcome: The Treatment Credibility/Expectancy Questionnaire
Description: The Treatment Credibility/Expectancy Questionnaire is composed of 4 questions that assess treatment credibility, or the extent to which a treatment seems logical and able to address patient complaints. The credibility scores may range from 4 to 36, with higher scores indicating greater endorsement of credibility.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | painTRAINER Pain Management Web Application
Number analyzed (Participants) | 21
score on a scale | 21 (5.6)

3. Secondary Outcome: Patient Pain: Change in Graded Chronic Pain Scale Characteristic Pain Intensity (GCPS-CPI) Score
Description: Graded Chronic Pain Scale Characteristic Pain Intensity (GCPS-CPI) score: GCPS-CPI is made up of 3 questions asking the patient to rate their pain Now, at its worst, and on average over the past 30 days. Scores on the index may range from 0 to 30, with higher scores indicative of greater characteristic pain. Outcome is measured in change from baseline.
Time Frame: baseline to 3 months after treatment
Measure: Mean (Standard Deviation); unit: score on a scale: decrease in pain score
Arm/Group | painTRAINER Pain Management Web Application
Number analyzed (Participants) | 21
score on a scale: decrease in pain score | 1.7 (2.0)

ADVERSE EVENTS:
Time Frame: Up to 12 weeks from baseline
Arm/Group | painTRAINER Pain Management Web Application
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/70/NCT05862870/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/70/NCT05862870/ICF_001.pdf